CLINICAL TRIAL: NCT04311372
Title: Sleep Wellness Program - University REST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID 2020 pandemic, was unable to get started
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, MICHAEL A GRANDNER, Associate Professor of Psychiatry, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TBD3
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2020-03

CONDITIONS: Poor Quality Sleep; Sleep Disturbance
Keywords: Mental Health; College Students; Sleep; Educational Intervention
MeSH Terms: conditions — Parasomnias; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: N=100 participants will be randomized to one of two groups.
  Group 1 | n =50 participants (Educational Session + Material from Educational Session (Handout form) + Access to Online Video Library)
  Group 2 | n =50 participants (Educational Session + Material from Educational Session (Handout form) ONLY)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educational session+Material+Videos (Group 1) (Experimental): n =50 participants (Educational Session + Material from Educational Session (Handout form) + Access to Online Video Library)
  Interventions: Behavioral: Educational Sesssion+Material+Videos
- Educational session+Material ONLY (Group 2) (Active Comparator): n =50 participants (Educational Session + Material from Educational Session (Handout form) ONLY)
  Interventions: Behavioral: Educational Sesssion+Material ONLY

INTERVENTIONS:
Behavioral: Educational Sesssion+Material+Videos — n =50 participants (Educational Session + Material from Educational Session (Handout form) + Access to Online Video Library)
  Other Names: Group 1
  Arms: Educational session+Material+Videos (Group 1)
Behavioral: Educational Sesssion+Material ONLY — n =50 participants (Educational Session + Material from Educational Session (Handout form) ONLY)
  Other Names: Group 2
  Arms: Educational session+Material ONLY (Group 2)

SUMMARY:
This study study aims to examine relationships between sleep and mental health and well-being among a more heterogeneous sample of students and apply the REST intervention to this group to determine whether we can improve sleep in this group and whether changes in sleep are associated with improvements in mental health.

DETAILED DESCRIPTION:
Poor mental health is a major problem among college students. Data from the World Health Organization (WHO) reports that 20% of college students likely meet criteria for a mental health condition, yet only approximately 16% of those with conditions received treatment. Data from the 2015 National College Health Assessment (N=67,308 from 108 colleges/universities) showed that 25% of the sample had a diagnostic history of a psychiatric condition. Further, this study found high rates of the presence of mental health symptoms in the past 12 months among students, with 35% reporting depression that interfered with functioning, 39% reporting overwhelming anger, 50% reporting hopelessness, 58% reporting overwhelming anxiety, 61% reporting loneliness, 66% reporting feeling very sad, 83% reporting exhaustion, and 87% reporting feeling overwhelmed. Self-harm was reported by 7% and 10% reported that they "seriously considered suicide."

Many previous studies have shown that sleep is strongly related to mental health, especially among your adults. In particular, our preliminary data from the 2011-2014 National College Health Assessment data show that each night of reported insufficient sleep was associated with an increased likelihood of also reporting hopelessness (28% increase per night of insufficient sleep), feeling overwhelmed (24%), exhaustion (31%), loneliness (21%), sadness (21%), functional problems (30%), anxiety (28%), anger (27%), desire to hurt self (21%), suicide ideation (30%), and suicide attempts (12%). In looking at UA students, we previously found that among student athletes, sleep is related to mental health. Sleep duration, sleep quality, insomnia, fatigue, and symptoms of sleep disordered breathing were all independently associated with depression, anxiety, and mental well-being.

In our previous work, we developed an intervention called "REST" (Recovery Enhancement and Seep Training) that was deployed among student athletes. This intervention included education, sleep tracking, a financial incentive (lottery system), and support. It was effective at increasing sleep duration (by M=77 mins) and improving sleep quality (increased sleep efficiency, reduced insomnia severity, and reduced fatigue). The present study aims to examine relationships between sleep and mental health and well-being among a more heterogeneous sample of students and apply the REST intervention to this group to determine whether we can improve sleep in this group and whether changes in sleep are associated with improvements in mental health.

ELIGIBILITY:
Inclusion Criteria:

* at least a score of 3 on the Pittsburgh Sleep Quality Index (indicating at least a minor problem with sleep quality).
* a score of at least 6 on the Epworth Sleepiness Scale (indicating at least moderate sleepiness).
* a score of at least 7 on the Insomnia Severity Index (indicating at least mild insomnia), or habitual sleep duration of less than 6 hours per night (indicating insufficient sleep).

Exclusion Criteria:

* score less than a 3 on the Pittsburgh Sleep Quality Index.
* score less than a 6 on the Epworth Sleepiness Scale.
* score less than a 7 on the Insomnia Severity Index.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Insomnia Severity Index (ISI) | Change from baseline to post-intervention, around 8 weeks after baseline
  The Insomnia Severity Index is a brief screening assessment tool designed to evaluate insomnia. Time frame: past 2 weeks. Measuring 7 items. Scores range from 0-28. Scores interpret as follow: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28). The higher the result, the more severe the insomnia is.
Changes in the Pittsburgh Sleep Quality Index (PSQI) | Change from baseline to post-intervention, around 8 weeks after baseline
  A subjective measure of sleep. Score ranges from 0-21. Higher scores indicate worse sleep quality.
Changes in the Fatigue Severity Scale (FSS) | Change from baseline to post-intervention, around 8 weeks after baseline
  The Fatigue Severity Scale is a self-reported scale measuring fatigue. Time frame: previous week. Measuring 9 items. Scores ranges from 9-63. Levels of fatigue interpret as follow: not suffering from fatigue (<36); presence of fatigue (>36). The higher the score, the greater fatigue is perceived.
Changes in the Epworth Sleepiness Scale (ESS) | Change from baseline to post-intervention, around 8 weeks after baseline
  The Epworth Sleepiness Scale is a self-administered questionnaire that's routinely used to assess daytime sleepiness. Time frame: previous 2 weeks. Measuring 8 items. Score ranges from 0-24. The higher the score, the higher average sleep propensity in daily life (ASP) or daytime sleepiness is.
Changes in the Assessment of Sleep Environment (ASE) | Change from baseline to post-intervention, around 8 weeks after baseline
  A questionnaire that measures the degree to which the physical environment disturbs sleep. It contains 13 items with scores ranging from 0-Strongly Disagree to 3-Strongly Agree. Higher scores suggest less optimal sleep environment.
Changes in the Center for Epidemiologic Studies Depression Scale (CES-D) | Change from baseline to post-intervention, around 8 weeks after baseline
  A short self-report scale designed to measure depressive symptomatology. Time frame: previous week. Measuring 20 items comprising 6 scales. Score ranges from 0-60. The higher the score is the greater the presence of depressive symptomatology.
Changes in the Patient Health Questionnaire (PHQ-9) | Change from baseline to post-intervention, around 8 weeks after baseline
  A self-administered questionnaire for common mental disorders, specifically in to the depression module. Time frame: past 2 weeks. Measuring 9 items. Scores ranges from 0-27. Levels of depression measure as follow: minimal (0-4); mild (5-9); moderate (10-14); moderately severe (15-19); severe (20-27).
Changes in Generalized Anxiety Disorder (GAD-7) | Change from baseline to post-intervention, around 8 weeks after baseline
  A brief self-report scale to identify probable cases of generalized anxiety. Time frame: past 2 weeks. Measuring 7 items. Scores ranges from 0-21. Levels of anxiety measure as follow: mild (0-9); moderate (10-14); severe (>15). The higher the score the greater presence of generalized anxiety.
Changes in Perceived Stress Scale (PSS) | Change from baseline to post-intervention, around 8 weeks after baseline
  A subjective scale measuring perceived stress. Measuring 10 items. Time frame: previous month. Score ranges from 0-40. Levels of stress measure as follow: low stress (0-13); moderate stress (14-26); high perceived stress (27-40). The higher the score, the greater stress is perceived.

SECONDARY OUTCOMES:
National College Health Assessment (NCHA) Mental Health Item | Change from baseline to post-intervention, around 8 weeks after baseline
  The NCHA Mental Health Item contains two brief questions regarding adapting after changes/hardships occur. The scores range from 0-Not at all true to 4-True all the time. A higher score equates to greater ability to adapt after changes.
Columbia Suicide Severity Rating Scale | Change from baseline to post-intervention, around 8 weeks after baseline
  The Columbia Suicide Severity Rating Scale (CSSRS) is a scale containing 16 items which measures suicidality in 3 distinct sections: severity, intensity, and behavior. Answers are "yes" or "no", and scores are determined based on yes/no responses to each question and an added sum of intensity of ideation, ranging from 2-25 with higher scores meaning more intense suicide ideation.
World Health Organization (WHO) Performance Questionnaire Item A9 | Change from baseline to post-intervention, around 8 weeks after baseline